CLINICAL TRIAL: NCT02110914
Title: Coach to Cope. Coaching Young Adults With Cystic Fibrosis - a Feasibility Study
Brief Title: A Coaching Intervention to Young Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Karin Bæk Knudsen, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-2-2013-FSP01
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis
Keywords: Feasibility study; Coaching; Health related quality of life; Adherence
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaching (Experimental): 10 coaching sessions over a period of 6 - 9 months. The intervention is life coaching based on principles of the co-active coaching model.
  Interventions: Behavioral: Coaching
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Coaching — Coaching is based on the principles of the Co-active coaching model and performed by a certified coach. At the first coaching session the coach and client will make an agreement about the format for subsequent coaching sessions. The first and the last coaching session will always be "face to face" at the hospital and last 1- 1½ hours. Intervening coaching sessions will be approximately 60 minutes by phone or face to face. In total, ten coaching sessions will be offered, one every 1-2 weeks early in the program and one every 2-4 weeks later in the process. The duration of the coaching intervention will be between 6 and 9 months.
  Other Names: Life coaching
  Arms: Coaching

SUMMARY:
The treatment burden for patients with cystic fibrosis (CF) is significant and poor adherence has been well-documented. The investigators hypothesize that a coaching intervention will empower young adults with CF to manage their lives with CF and improve health-related quality of life (HRQoL). The main aim of the study is to establish the feasibility and acceptability of a life-coaching intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic fibrosis (CF), confirmed by clinical findings, identification of two disease-causing CF- mutations, and a positive sweat test
* Patient at the Copenhagen CF Centre

Exclusion Criteria:

* Severe intellectual impairment or insufficient mastery of the Danish language, determined by incapacity to independently complete the questionnaires

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | 12 months
  Willingness of eligible participants to be recruited and randomized, adherence to the intervention and attrition rates

SECONDARY OUTCOMES:
Health Related Quality of Life | Up to 21 months
  The primary effect outcome is change in health-related quality of life (HRQoL), with special focus on the two domains: Social and Emotional functioning on the Cystic Fibrosis Questionnaire-Revised (CFQ-R).
  For the intervention group HRQoL is measured at baseline, midway (after 5 coaching sessions), post intervention (after 10 coaching sessions) and at follow up (12 months post intervention) For the control group HRQoL is measured at baseline, midway (after 4 months), post intervention (after 9 months) and at follow up (12 months post intervention)
Self-reported Adherence | 21 months
  Morisky Medication Adherence Scale (MMAS-8), questionnaires are completed at baseline, and 4, 9 and 21 months after baseline
Pharmacy Refill Histories | up to 1 year
  Data from the pharmacy database will be collected for two four- month periods: four months prior to the intervention and four months at the end of the intervention. The last four months will be two months prior to end of study and two months after for the intervention group, and seven to eleven month after baseline for the control group
Self-efficacy | 21 month
  General Self-Efficacy Scale (GSE), questionnaires are completed at baseline, and 4, 9 and 21 months after baseline
Clinical data | 21 months
  Lung function test (spirometry, FEV1), Body Mass Index (BMI) and Hemoglobin A1C (HbA1C), Data will be collected from the medical chart at baseline, and 4, 9 and 21 months after baseline

OTHER OUTCOMES:
The participants' experiences with and acceptability of the intervention | 12 month
  In depth interviews with participants from the intervention arm after their last coaching session

CONTACTS AND LOCATIONS:
Overall Officials: Laust H Mortensen, PhD, Study Chair — Department of Public Health at the University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark